CLINICAL TRIAL: NCT03432481
Title: Open-Label Investigational Testing of Bodycad Unicompartmental Knee Prosthesis (UKS) in Human Subjects With Medial Unicompartmental Knee Osteoarthritis
Brief Title: Investigational Testing of Bodycad Unicompartmental Knee Prosthesis (UKS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interruption due to the ongoing corporate restructuring, which has resulted in the cessation of our interest in
  pursuing any clinical activities related to the product.
Sponsor: Laboratoires Bodycad Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-PB001-42
Record Dates: First submitted 2018-01-22; First posted 2018-02-14 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Knee Arthroplasty using BUKS (Experimental): Unicompartmental Knee Arthroplasty Surgery
  Interventions: Procedure: Unicompartmental Knee Arthroplasty Surgery; Device: Bodycad Unicompartmental Knee System (BUKS)

INTERVENTIONS:
Procedure: Unicompartmental Knee Arthroplasty Surgery — Unicompartmental Knee Arthroplasty Surgery using the Bodycad Unicompartmental Knee System (BUKS)
Device: Bodycad Unicompartmental Knee System (BUKS) — Unicompartmental Knee Arthroplasty Surgery using the Bodycad Unicompartmental Knee System (BUKS)

SUMMARY:
This study is designed to observe clinical outcomes of patient-specific knee arthroplasty in patients with osteoarthritis of the medial condyle.

DETAILED DESCRIPTION:
The patient-specific Bodycad Unicompartmental Knee System will be implanted on patients with knee osteoarthritis of the medial condyle. The study's hypothesis is that personalized shape and fit of patient-specific knee replacement prosthesis will provide a greater stability and a more natural knee motion in addition to a faster recovery when compared to traditional knee replacement systems. This study is designed to provide a five-years follow-up clinical data on safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Medial unicompartmental knee osteoarthritic disease diagnosed on the basis of the American College of Rheumatology criterion with radiographic confirmation (Kellgren- Lawrence grade 3 or higher, on a scale of 0 to 4, with higher numbers indicating more severe signs of osteoarthritis); or isolated medial compartment post-traumatic arthritis supported by long film (x-ray);
2. Between the ages of at least 45 years and 70 years (inclusive) at the time of enrollment;
3. Stable health as judged by the Investigator;
4. Willingness to adhere to the protocol requirements as evidenced by the informed consent form duly read, signed and dated by the subject.

Exclusion Criteria:

1. Presence of active or latent infection in the knee;
2. Diagnosis of rheumatoid arthritis or avascular necrosis;
3. Presence of moderate patellofemoral osteoarthritic disease or patellofemoral maltracking;
4. Anterior or posterior translational, varus or valgus ligamentous knee instability and/or deformity;
5. Extension deficit > 15˚ of affected knee;
6. History of ligament surgery on the affected knee, patient that already have a prosthesis on other condyles of the affected knee and/or patient requiring a revision knee replacement surgery;
7. History of proximal tibial fracture, non-union, deformity or oblique joint line;
8. Deficient bone mass that may not provide adequate support and / or fixation;
9. Skeletal immaturity;
10. Obesity: BMI above 35
11. Risk of exposing the prosthesis to overload by the practice of contact or high impact sports such as: baseball, hockey, basketball, football, soccer, karate, skiing etc;
12. Known sensitivity to CoCrMo, Titanium, and polyethylene components of the UKS Prosthesis used in the manufacturing of the prosthesis;
13. Pre-existing medical conditions such as history of cancer other than skin cancer, poorly controlled diabetes, systemic infections, immunocompromised, fibromyalgia or other general body pain conditions, which, in the opinion of the Investigator, interfere with the conduct of the study;
14. Neuromuscular condition that could lead to an unacceptable risk of instability of the prosthesis or other postoperative complications;
15. Subjects, in the opinion of the Investigator, who are unlikely to comply with the protocol (e.g. active alcoholism, drug dependency or psychotic state, unable or unwilling to adhere to study visit schedule);
16. Pregnant or nursing female subjects; or female subjects planning on becoming pregnant within the next 60 months from enrollment;
17. Subjects under guardianship, hospitalized in a public or private institution, for a reason other than research, or subject deprived of freedom;
18. Participation in an active stage of any drug, intervention or treatment trial within 30 days of enrollment.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Knee Society Score (KSS) Objective | Baseline, post-operative months 3, 6, 12, 24, 36, 48 and 60
  Assessment of improvement of clinical outcomes following BUKS implantation using the KSS questionnaire, to evaluate the clinical performance of the articulation
Change from baseline in Knee Osteoarthritis Outcome Score (KOOS) | Baseline, post-operative months 3, 6, 12, 24, 36, 48 and 60
  Assessment of improvement of activity levels following BUKS implantation surgery using the KOOS questionnaire

SECONDARY OUTCOMES:
Change from baseline in mechanical axis measurement. | Baseline and post operative week 1
  Determine by radiographic analysis Varus or Valgus, expected value are +/- 3 degrees
Change from baseline of implant position fixation | Post operative week 6, months 6, 12, 24, 36, 48 and 60
  The anteroposterior and medial lateral slop will be evaluated according to initial planed position. The measured angles will be compared with initial planning. The expected values are +/- 1.5 degree.
Change from baseline on bone loss and cementation | Post operative week 6, months 6, 12, 24, 36, 48 and 60
  Those measurements will be done on x-ray of the patient joint following Knee Society Radiological evaluation form.The tibial component acceptable score for this device will be 2.5 mm. The femoral component acceptable score for this device will be 6 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Belzile, MD, Principal Investigator — CHU de Quebec - Hopital de l'Enfant-Jésus; Brian Hamlin, MD, Study Chair — Renaissance Orthopedics; Geoffroy Rivet-Sabourin, PhD, Study Director — Laboratoires Bodycad Inc.
Locations (1):
- CHU de Quebec - Universite Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided